CLINICAL TRIAL: NCT00916097
Title: A Multicenter Phase II Trial of Docetaxel Combined With Cisplatin (CDDP) as a Neo-Adjuvant Chemotherapy in Patients With Loco Regionally Advanced Undifferentiated Carcinoma of Nasopharyngeal Type (UCNT)
Brief Title: NPC Study : TAX + CIS Neoadjuvant in Patients With Loco Regionally Advanced Undifferentiated Carcinoma of Nasopharyngeal Type (UCNT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976F_2502
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

ARMS (1):
- 1 (Experimental): docetaxel 75mg/m2 in combination with cisplatin 75mg/m2 given every 3 weeks for 3 cycles
  Interventions: Drug: DOCETAXEL(XRP6976)

INTERVENTIONS:
Drug: DOCETAXEL(XRP6976) — docetaxel 75mg/m2 by intravenous infusion over 60 minutes on Day 1 of a 3-week cycle

SUMMARY:
Primary Objective:

To estimate the overall response rate after neo-adjuvant chemotherapy of Docetaxel 75 mg/m2 in combination with Cisplatin 75 mg/m2 given for 3 cycles, and followed by conventional radiotherapy in UCNT.

Secondary Objectives:

To evaluate:

* The radiological response after chemotherapy and radiotherapy
* The pathological response after chemotherapy by cavum biopsy

To estimate:

* The duration of overall response
* The time to progression (T.T.P)

To analyze:

* The overall survival
* The safety profile

ELIGIBILITY:
Inclusion criteria:

* Written or witnessed oral informed consent prior to beginning specific protocol procedures >Histologically proven undifferentiated carcinoma of nasopharyngeal type (UCNT- stage II-III OMS) at first diagnosis
* Staging of disease: stage III, IV A, IV B (UICC/AJCC, 1997 classification), any T, N2 - N3 UCNT, without metastasis
* Adenopathy > 3 cm
* Patients are required to have an unidimensionally measurable disease with RECIST method
* Performance status 1 or karnofsky index 3
* Previous therapy: Chemotherapy :none Radiation therapy: none Surgery: none
* Laboratory requirements

Exclusion criteria:

* Prior chemotherapy or / and radiotherapy
* Metastatic disease (M as per the UCCI/AJC classification)
* Past or current history of neoplasm other than UCNT, except for curatively treated non melanoma skin cancer or in situ carcinoma of the cervix or other cancer,curatively treated and with no evidence of disease at the previous 5 years
* Pregnant, or lacting, patients of childbearing potential must implement adequate contraceptive measures during study participation
* Pre-existing motor or sensory neurotoxicity of a severity 3 grade 2 according to NCI criteria
* Others serious illness or medical condition:

  1.Congestive heart failure or unstable angina pectoris even if it is medically controlled 2.Previous history of myocardial infraction within 1 year from study entry 3.Uncontrolled hypertension or high risk uncontrolled arrhythmias 4.Uncontrolled peptic ulcer, unstable diabetes mellitus susceptible to contraindicate any use of corticoids 5.Concomitant treatment with corticoids initiated > 6 months prior to study entry is given to the dose of methylprednisolone or equivalent 3 20 mg 6.Definite contraindications for the use of Corticoids 7.Concurrent treatment with other experimental drugs 8.Participation in another clinical with any investigational drug within 30 days prior to study entry 9.Performance status = 2,3,4 or karnofsky index < 80 10. History of significant neurologic or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2002-07; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of tumor response in patients with measurable disease according to RECIST criteria | on day 21 of each treatment cycle for neoadjuvant chemotherapy, on day 64 and day 71 (3 to 4 weeks after the third chemotherapy)

SECONDARY OUTCOMES:
Evaluation of the radiological response after chemotherapy and radiotherapy | from baseline to the end of the study
Evaluation of the pathological response after chemotherapy | between day 64 and day 71 of the treatment
Overall response duration | from baseline to the end of the study
Estimation of the time to progression | from baseline to the end of the study
Overall survival | from baseline to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Christian Fassotte, Study Director — Sanofi
Locations (3):
- Sanofi-Aventis Administrative Office, Algiers, Algeria
- Sanofi-Aventis Administrative Office, Casablanca, Morocco
- Sanofi-Aventis Administrative Office, Mégrine, Tunisia